CLINICAL TRIAL: NCT04257656
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Remdesivir in Hospitalized Adult Patients With Severe COVID-19.
Brief Title: A Trial of Remdesivir in Adults With Severe COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The epidemic of COVID-19 has been controlled well in China, no eligible patients can be enrolled at present.
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-China remdesivir 2
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Remdesivir; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remdesivir group (Experimental): active remdesivir
  Interventions: Drug: Remdesivir
- Control group (Placebo Comparator): Placebos matched remdesivir
  Interventions: Drug: Remdesivir placebo

INTERVENTIONS:
Drug: Remdesivir — RDV 200 mg loading dose on day 1 is given, followed by 100 mg iv once-daily maintenance doses for 9 days.
  Other Names: GS-5734
  Arms: Remdesivir group
Drug: Remdesivir placebo — RDV placebo 200 mg loading dose on day 1 is given, followed by 100 mg iv once-daily maintenance doses for 9 days.
  Arms: Control group

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (SARS-CoV-2) from these pneumonia patients and developed a real-time reverse transcription PCR (real-time RT-PCR) diagnostic assay.

Given no specific antiviral therapy for COVID-19 and the ready availability of remdesvir as a potential antiviral agent, based on pre-clinical studies in SARS-CoV and MERS-CoV infections, this randomized, controlled, double blind trial will evaluate the efficacy and safety of remdesivir in patients hospitalized with severe COVID-19.

DETAILED DESCRIPTION:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (SARS-CoV-2) from these pneumonia patients and developed a real-time reverse transcription PCR (real-time RT-PCR) diagnostic assay.

Whilst the outbreak is likely to have started from a zoonotic transmission event associated with a large seafood market that also traded in live wild animals, it soon became clear that person-to-person transmission was also occurring. The number of cases of infection with COVID-19 identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally. Mathematical models of the expansion phase of the epidemic suggested that sustained person-to-person transmission is occurring, and the R-zero is substantially above 1, the level required for a self-sustaining epidemic in human populations.

The clinical spectrum of COVID-19 illness appears to be wide, encompassing asymptomatic infection, a mild upper respiratory tract infection, and severe viral pneumonia with respiratory failure and even death. Although the per infection risk of severe disease remains to be determined, case-fatality risk of 11-14% has been reported in several initial studies of seriously ill patients and case-fatality has been estimated approximately at 2% overall. Also the large number of cases in Wuhan has resulted in a large number of patients hospitalised with pneumonia requiring supplemental oxygen and sometimes more advance ventilator support.

This new coronavirus, and previous experiences with SARS and MERS-CoV, highlight the need for therapeutics for human coronavirus infections that can improve clinical outcomes, speed recovery, and reduce the requirements for intensive supportive care and prolonged hospitalisation.

Given no specific antiviral therapy for COVID-19 and the ready availability of remdesvir as a potential antiviral agent, based on pre-clinical studies in SARS-CoV and MERS-CoV infections, this randomized, controlled, double blind trial will evaluate the efficacy and safety of remdesivir in patients hospitalized with severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of signing Informed Consent Form
2. Laboratory (RT-PCR) confirmed COVID-19.
3. Lung involvement confirmed with chest imaging
4. Hospitalized with a SaO2/SPO2≤94% on room air or Pa02/Fi02 ratio <300mgHg
5. ≤12 days since illness onset
6. Willingness of study participant to accept randomization to any assigned treatment arm.
7. Must agree not to enroll in another study of an investigational agent prior to completion of Day 28 of study.

Exclusion Criteria:

1. Physician makes a decision that trial involvement is not in patients' best interest, or any condition that does not allow the protocol to be followed safely.
2. Severe liver disease (e.g. Child Pugh score ≥ C, AST>5 times upper limit)
3. Pregnant or breastfeeding, or positive pregnancy test in a predose examination
4. Patients with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
5. Will be transferred to another hospital which is not the study site within 72 hours.
6. Receipt of any experimental treatment for COVID-19 within the 30 days prior to the time of the screening evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Improvement (TTCI) [Censored at Day 28] | up to 28 days
  The primary endpoint is time to clinical improvement (censored at Day 28), defined as the time (in days) from randomization of study treatment (remdesivir or placebo) until a decline of two categories on a six-category ordinal scale of clinical status (1 ꞊ discharged; 6 ꞊ death) or live discharge from hospital.
  Six-category ordinal scale:
  6. Death; 5. ICU, requiring ECMO and/or IMV; 4. ICU/hospitalization, requiring NIV/ HFNC therapy; 3. Hospitalization, requiring supplemental oxygen (but not NIV/ HFNC); 2. Hospitalization, not requiring supplemental oxygen;
  1. Hospital discharge or meet discharge criteria (discharge criteria are defined as clinical recovery, i.e. fever, respiratory rate, oxygen saturation return to normal, and cough relief).
  Abbreviation: IMV, invasive mechanical ventilation; NIV, non-invasive mechanical ventilation; HFNC, High-flow nasal cannula.

SECONDARY OUTCOMES:
Clinical status | days 7, 14, 21, and 28
  Clinical status, assessed by the ordinal scale at fixed time points (days 7, 14, 21, and 28).
Time to Hospital Discharge OR NEWS2 (National Early Warning Score 2) of ≤ 2 maintained for 24 hours. | up to 28 days
  Time to Hospital Discharge OR NEWS2 (National Early Warning Score 2) of ≤ 2 maintained for 24 hours.
All cause mortality | up to 28 days
Duration (days) of mechanical ventilation | up to 28 days
Duration (days) of extracorporeal membrane oxygenation | up to 28 days
Duration (days) of supplemental oxygenation | up to 28 days
Length of hospital stay (days) | up to 28 days
Time to 2019-nCoV RT-PCR negativity in upper and lower respiratory tract specimens | up to 28 days
Change (reduction) in 2019-nCoV viral load in upper and lower respiratory tract specimens as assessed by area under viral load curve. | up to 28 days
Frequency of serious adverse drug events | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bin Cao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582
- [Derived] Wang Y, Zhou F, Zhang D, Zhao J, Du R, Hu Y, Cheng Z, Gao L, Jin Y, Luo G, Fu S, Lu Q, Du G, Wang K, Lu Y, Fan G, Zhang Y, Liu Y, Ruan S, Liu W, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Evaluation of the efficacy and safety of intravenous remdesivir in adult patients with severe COVID-19: study protocol for a phase 3 randomized, double-blind, placebo-controlled, multicentre trial. Trials. 2020 May 24;21(1):422. doi: 10.1186/s13063-020-04352-9. PMID 32448345
- [Derived] Wang Y, Zhang D, Du G, Du R, Zhao J, Jin Y, Fu S, Gao L, Cheng Z, Lu Q, Hu Y, Luo G, Wang K, Lu Y, Li H, Wang S, Ruan S, Yang C, Mei C, Wang Y, Ding D, Wu F, Tang X, Ye X, Ye Y, Liu B, Yang J, Yin W, Wang A, Fan G, Zhou F, Liu Z, Gu X, Xu J, Shang L, Zhang Y, Cao L, Guo T, Wan Y, Qin H, Jiang Y, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Remdesivir in adults with severe COVID-19: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2020 May 16;395(10236):1569-1578. doi: 10.1016/S0140-6736(20)31022-9. Epub 2020 Apr 29. PMID 32423584